CLINICAL TRIAL: NCT04630366
Title: A Phase 1, First Time in Man Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of NST-1024 in Healthy Subjects and Otherwise Healthy Subjects With Elevated Triglycerides
Brief Title: A Phase 1, First Time in Humans Study of NST-1024
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NorthSea Therapeutics B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NST-1024-01
Record Dates: First submitted 2020-11-05; First posted 2020-11-16 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NST-1024 (Experimental): NST-1024 capsules given once daily for up to 14 days
  Interventions: Drug: NST-1024
- Placebo (Placebo Comparator): Matching placebo capsules to NST-1024 given once daily for up to 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NST-1024 — NST-1024
  Arms: NST-1024
Drug: Placebo — Matching placebo to NST-1024
  Arms: Placebo

SUMMARY:
A first time in man study of NST-1024

DETAILED DESCRIPTION:
A Phase 1, First Time in Man Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of NST-1024 in Healthy Subjects and Otherwise Healthy Subjects with Elevated Triglycerides. This will be a double-blind, randomised, placebo-controlled, single and multiple oral dose study conducted in 2 parts. In part A up to 6 cohorts of 8 healthy volunteers will receive single ascending doses of NST-1024 or matching placebo. I part B up to 4 cohorts of 10 otherwise healthy volunteers, with elevated triglycerides will receive daily multiple ascending doses of NST-1024 for 14 days

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-32 kg/m2
* In good health
* Females will not be pregnant or lactating. Females of childbearing potential must agree to use contraception
* Male subjects must agree to use contraception and refrain from donation of sperm
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
* Subjects must have TG levels > 150 mg/dL at screening (Part B only).

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, CV, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
* Aspartate aminotransferase, ALT, GGT, ALP, or total bilirubin > 1.2 × ULN at Screening or (first) Check-in, confirmed by 1 repeat if necessary
* History of alcoholism or drug/chemical abuse within 2 years prior to Check-in.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days or 5 half-lives (whichever is longer) prior to dosing.
* Use of tobacco- or nicotine-containing products within 1 month prior to Screening, or positive cotinine test at Screening or Check-in.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 4 weeks
  incidence and severity of adverse events

SECONDARY OUTCOMES:
AUC | 3-17 days
  Area under the PK curve
Cmax | 3-17 days
  Maximum plasma concentration
Half life | 3-17 days
  time to reduction in plasma levels by 50%

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Leeds Clinical Research Unit, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No